CLINICAL TRIAL: NCT03772808
Title: Effects of LycoComfort™ Supplementation on Symptoms Associated With Lower Urinary Tract Symptoms (LUTS)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: LycoRed Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: OBVIO-LYC-001
Record Dates: First submitted 2018-11-19; First posted 2018-12-11 (Actual); Last update posted 2019-07-02 (Actual); Status verified 2019-06

CONDITIONS: BPH; Lower Urinary Tract Symptoms
MeSH Terms: conditions — Lower Urinary Tract Symptoms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Lycocomfort (Experimental): The once-daily supplement LycoComfort™ is a combination of lycopene and beta-sitosterol, a chemically defined extract of phytosterols with beta-sitosterol as the main component,
  Interventions: Dietary Supplement: Lycocomfort

INTERVENTIONS:
Dietary Supplement: Lycocomfort — Evaluate of the perceived efficacy of LycoComfort™ supplements in alleviating symptoms associated with lower urinary tract symptoms (LUTS) and general prostate discomfort over the duration of 12 weeks intervention

SUMMARY:
This study will evaluate LycoComfort™ supplementation in alleviating symptoms associated with LUTS, BPH, and general prostate concerns.

Inflammation, oxidative stress and androgenic activity in the prostate are proven catalysts of BPH, ultimately leading to increased prostate cell proliferation. The once-daily supplement LycoComfort™, will be under investigation for symptom relief and will be taken by participants for a duration of 12 weeks.

DETAILED DESCRIPTION:
LycoComfort™ is a dietary supplement containing tomato extract and phytosterols, ingredients that have been associated with relief of symptoms associated with general prostate discomfort and Lower Urinary Tract Symptoms (LUTS).

The purpose of this study is to evaluate changes in these symptoms after taking this supplement daily for 12 weeks.

Although it was not until the latter part of the twenties century that investigators began to explore the importance of lycopene, the benefits of this natural carotenoid are well studied. A number of clinical trials have shown lycopene to be effectual for alleviating prostate discomfort, symptoms of BPH and LUTS.

The American Urological Association estimates that 90% of men between 45 and 80 years of age suffer some symptoms of LUTS. Several pathophysiological mechanisms are believed to lead to LUTS and BPH, including oxidative damage, inflammation and sympathetic nervous system issues. High blood lycopene concentrations have been suggested in epidemiological trials to be associated with decreases in oxidative stress and contributions to disease prevention overall. Also, clinical trials have shown that higher levels of lycopene in the blood are associated with a reduced risk of prostate cancer, as well as other inflammatory conditions.

ELIGIBILITY:
Inclusion Criteria:

* Males, age 40 and older
* A score of 8 or greater on a self-administered I-PSS test

Exclusion Criteria:

* Acute or chronic prostatitis
* Acute urinary retention
* Allergy or sensitivity to any of the test product components (tomato [lycopene] or beta-sitosterol)
* Cancer of the prostate (PCa) or other cancers, current or a history of PCa
* Chronic diseases of the kidneys and/or liver
* Hematuria of unknown etiology
* Infection or malfunction of the urinary tract
* Inflammatory diseases of the urogenital tract
* Medication, herbal supplementation or other substance use for the treatment of urinary symptoms, BPH/LUTS, or erectile dysfunction, including medications which may affect hormonal status within 30 days before screening. These may include, but are not limited to: Sildenafil/Viagra; Tadalafil/Cialis; Vardenafil/Levitra; "Herbal Viagra"; Alpha-Blockers; Oral Steroids, Spironolactone or Testosterone
* Previous radiotherapy of prostate
* Previous surgery of the prostate, bladder or urethra

Min Age: 40 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2018-11-16 (Actual); Primary Completion 2019-04-30 (Actual); Study Completion 2019-06-15 (Actual)

PRIMARY OUTCOMES:
Number of patients with a change in International Prostate Symptom Score (I-PSS) | Enrollment to 12 weeks
  Change from enrollment to week 12 in prostate symptoms, measured by the Prostate Symptom Score questionnaire (I-PSS) ranged 1-35 points (1-7: Mild 8-19: Moderate 20-35: Severe).

SECONDARY OUTCOMES:
Number of patients with a significant improvement in International Prostate Symptom Score (I-PSS) | 12 weeks
  The number of subjects with a clinically significant improvement in International Prostate Symptom Score (I-PSS) at week 12, defined as an improvement of at least 3 points in a 1-35 point scale.
Number of patients with a change in Core Lower Urinary Tract Symptom Score (CLSS) | 12 weeks
  Change from enrollment to week 12 in urinary symptoms, measured by Core Lower Urinary Tract Symptom Score (CLSS), ranged 1-31 points.
Satisfaction from treatment evaluated by "User satisfaction questionnaire" | 12 weeks
  Subject satisfaction with the LycoComfort™ supplement, as derived from responses to "User satisfaction Questionnaire" ( 5 point Likert scale, ranged 8-45 points).
Adverse events (AEs) | 12 weeks
  Adverse events (AEs) reported during the treatment period and classified by the Investigator as to intensity, relationship to study procedures, and seriousness

OTHER OUTCOMES:
Number of patients with a change in Brief Sexual Function Index (BSFI) score | 12 weeks
  Change from enrollment to week 12 in sexual function, measured by Brief Sexual Function Index (BSFI) score ( ranged 0-44 points)

CONTACTS AND LOCATIONS:
Overall Officials: Parth Shah, MD, Principal Investigator — ObvioHealth
Locations (1):
- Obvio Health, Orlando, Florida, United States

IPD SHARING:
Plan to Share IPD: No